CLINICAL TRIAL: NCT03495440
Title: Families of Youth with Developmental Disabilities: a Theory-Based Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1246
Record Dates: First submitted 2017-05-24; First posted 2018-04-12 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Family Conflict; Marital Conflict; Communication
Keywords: Emotional Security; Intellectual Disability; Developmental Disability
MeSH Terms: conditions — Communication; Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Center Sessions (Experimental): Treatment condition in which participants receive psychoeducation and communication coaching.
  Interventions: Behavioral: Center Sessions
- At-home (Active Comparator): Active, self-study control condition in which participants receive regular communication with study personnel and self-study materials to review on their own.
  Interventions: Behavioral: At-home

INTERVENTIONS:
Behavioral: Center Sessions — Program to support relationships and communication between parents and typically developing adolescent siblings of individuals with intellectual and/or developmental disabilities.
  Arms: Center Sessions
Behavioral: At-home — Self-study resources paired with regular contact with study personnel.
  Arms: At-home

SUMMARY:
This study is designed to evaluate a preventive intervention program designed to support families (parents and typically developing adolescent siblings) that include a child with an intellectual and/or developmental disability. Participant families will be randomly assigned to either the treatment condition, in which they will receive psychoeducation and communication coaching over a four-week period, or the control condition, in which they will receive self-study materials. All subjects will participate in a pre-test assessment and three post-test assessments over the course of the year.

DETAILED DESCRIPTION:
A critical need exists for an evidence-based program to ameliorate the impact of family stress and conflict on the overall well-being of parents and TD siblings, as well as individuals with IDD. Our objective in this study is to test the efficacy for parents, TD siblings, and children with IDD of an adaptation of the psycho-educational and communication training approach used in a previously validated prevention/intervention program for community families, and to examine the mechanisms associated with change processes that occur as a result of the 4-week program. Our long-term goal is to increase the availability and affordability of empirically-supported family-systems approaches to reduce family stress and conflict in families of individuals with IDD. Our central hypothesis is that participation in the program will support the identified needs of families with a child with IDD, improve the well-being and adjustment of parents, increase emotional security and adjustment for TD siblings, and be associated with improvements in adaptive functioning for individuals with IDD. This central hypothesis is supported by promising qualitative evidence and preliminary analyses from an ongoing pilot study using the adapted curriculum included in the present proposal. Our rationale is that providing a family-systems approach to improving the family environment will support the well-being of each family member, including the child with IDD. The specific aims are: (1) determining the efficacy of the program for parents, (2a) determining the efficacy of the program for typically developing siblings, (2b) testing process models, guided by the Emotional Security Theory (EST; Davies & Cummings, 1994), to explain how and why and for whom and when changes occur as a result of the program, and (3) examining the impact of the program on individuals with IDD. Families (n=150) that include a child with IDD and a TD sibling between 11 and 17 years of age, will be randomly assigned to one of two groups: (1) parent and typically developing sibling intervention, or (2) resource only control. Multi-method assessments of all family members will be obtained at pre- and post-intervention visits, and 6-month and 1-year follow-ups. The approach is innovative because it addresses multiple family members' needs, tests theory about explanatory models for program impact, and utilizes a brief, psycho-educational format and a RCT design to evaluate its efficacy. This research is significant because it will create an inexpensive model program for family-system-level interventions for families of children with IDD, benefiting parents, siblings and the child with IDD, including evaluations of program effectiveness in standing community centers.

ELIGIBILITY:
Inclusion Criteria:

* Participants in all conditions will include mothers, fathers, TD siblings between 11 and 17 years old, and individuals with IDD of any age.
* Participants must be able to understand and respond to survey questions in English
* Parents must be cohabitating, with both participating children living in their home.
* Individual with IDD falls into one or more of the following categories: 1) meets criteria for an intellectual disability, which would mean a measured IQ of 70-75 or lower and a measured Adaptive Functioning score of 70-75 or lower, 2) meets criteria for an Autism Spectrum Disorder based on an evaluation using the ADOS-2, SCQ, and expert clinical judgment based on DSM-5 ASD criteria, or 3) has a medically verified genetic condition (e.g., Down syndrome, Fragile X syndrome, Williams syndrome, Angelman syndrome, others) that is generally considered to be a developmental disability, and shows cognitive or adaptive functioning deficits (70-75 or below) although not necessarily deficits in both categories as would be needed for an Intellectual Disability diagnosis.

Exclusion Criteria:

* Siblings identified as typically developing will be excluded 1) with a score of 10 or higher on the SCQ-L, if a subsequent ADOS suggests that they have an ASD diagnosis, or 2) with a WASI-II score of 75 or lower.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in marital satisfaction -- Short Marital Adjustment Scale (SMAT) | 1 year
  15-item parent self-report questionnaire measuring indices of marital satisfaction, including matters of disagreement, relationship dynamics, and happiness.
Change in hostile interparental conflict -- O'Leary Porter Scales (OPS) | 1 year
  10-item parent self-report questionnaire designed to measure overt marital hostility exhibited in front of the children.
Change in family functioning -- Family Environment Scale (FES) | 1 year
  27-item self-report measure that assesses dimensions of family functioning, specifically, the social domain of family relationships (cohesion, expressiveness, and conflict) to be completed by parents and typically developing siblings.
Change in typically developing siblings' perception of interparental conflict -- Children's Perception of Inter-parental Conflict (CPIC) | 1 year
  19-item self-report questionnaire that captures three dimensions of marital conflict (frequency, intensity, and resolution) perceived by children.
Change in typically developing siblings' levels of attachment to parents -- Inventory of Parent and Peer Attachment (IPPA) | 1 year
  25-item self-report questionnaire designed to assess adolescents' perceptions of the positive and negative affective dimension of relationships with their parents and peers. Typically developing siblings complete two forms (father and mother) on three scales: trust, communication, and alienation.
Change in typically developing siblings' emotional security -- Security in the Subsystem (SIS) and Security in the Family System (SIFS) | 1 year
  The SIS is a child-report of the feelings and behaviors experienced when witnessing marital conflict. The SIFS is a self-report measure of adolescents' security in the family as a whole. Scores will be used in latent variables as a broad indicator of typically developing siblings' emotional security.
Change in typically developing siblings' adjustment -- Strengths and Difficulties Questionnaire (SDQ) | 1 year
  25-item parent-report measure of prosocial behavior and psychopathology in their children.
Change in typically developing siblings' behavior -- Youth Self-Report (YSR) | 1 year
  Adolescent self-report measure of perceived externalizing and internalizing behaviors.
Change in typically developing siblings' depressive symptomatology -- Child Depression Inventory (CDI) | 1 year
  27-item self-report questionnaire measuring the extent of depression symptoms in children.
Change on parents' depressive symptomatology - Beck Depression Inventory (BDI-II) | 1 year
  Parent self-report measure used to assess the severity of depression symptoms.
Change in parents' problem drinking behaviors -- Parental Alcohol Experiences scale (PAE) | 1 year
  Parent self-report measure that provides a continuous measure of parental problem drinking.
Change in the quality of family conflict interactions -- Family Interactions Coding System (FICS) | 1 year
  Video recorded quadratic (parent, TD sibling, child with IDD) interactions during which families discuss a topic of conflict are coded using an observational coding system to assess overall levels of constructiveness, destructiveness and resolution.
Change in the quality of couples' conflict interactions -- Family Interactions Coding System (FICS) | 1 year
  Video recorded dyadic (interparental) interactions during which couples discuss a topic of conflict are coded using an observational coding system to assess overall levels of constructiveness, destructiveness and resolution.
Change in family interactions in the home -- Daily Diaries | 6 months
  Parents complete 15 daily diaries following the 6-month and 12-month follow up assessments comprising of self-reports on the occurrence and quality of daily interparental and parent-child interactions.

SECONDARY OUTCOMES:
Change in adaptive functioning for individuals with IDD - Vineland Adaptive Behavior Scales II | 1 year
  Parent report measure describing skills and skill development in individuals with intellectual and/or developmental disabilities. Subscales focus on four domains: (1) Communication, (b) Daily Living Skills, (c) Socialization, and (d) Motor Skills. The domain composite scores make up the overall Adaptive Behavior Composite. The Internalizing and Externalizing subscales, and one subset of items labeled "Other" make up the optional Maladaptive Behavior Index. This index provides a measure of undesirable behaviors that may interfere with an individual's adaptive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Cummings, PhD, Principal Investigator — University of Notre Dame
Locations (2):
- United States (2):
  - Wm. J. Shaw Center for Children and Families, Fort Wayne, Indiana
  - Wm. J. Shaw Center for Children and Families, South Bend, Indiana

IPD SHARING:
Plan to Share IPD: No